CLINICAL TRIAL: NCT05701579
Title: Assessment of Anterior Cruciate Ligament (ACL) Degeneratio Mucosa Treatment
Status: Recruiting | Type: Observational
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Konrad Malinowski MD, Director of Artromedical Konrad Malinowski Clinic and Principal Investigator, Artromedical Konrad Malinowski Clinic
Other Study IDs: 1-pro-ar-2023
Record Dates: First submitted 2023-01-06; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ACL Degeneratio Mucosa: Patients with ACL Degeneratio Mucosa
  Interventions: Procedure: ACL "decompression"

INTERVENTIONS:
Procedure: ACL "decompression" — The technique of ACL "decompression" by the means of longitudinal incisions and evacuation of extrafibrous mucoid tissue.

SUMMARY:
Anterior Cruciate Ligament (ACL) Degeneratio Mucosa is a condition resulting from mucoid degeneration of ACL. Exact etiology is unknown, however ACL Degeneratio Mucosa impairs everyday functioning. In the literature there were some reports of treatment by ACL excision and subsequent reconstruction, however such treatment brings risk of deteriorated function. In this study the investigator will evaluate the technique of ACL "decompression" by the means of longitudinal incisions and evacuation of extrafibrous mucoid tissue.

ELIGIBILITY:
Inclusion Criteria:

* patients with ACL degeneratio mucosa decided to undergo a surgical treatment
* range of motion impairment caused by mucoid or cystic changes in ACL confirmed by MRI

Exclusion Criteria:

* non-adherence to the study protocol
* active knee inflammation
* range of motion impairment due to other extra- and intra-articular reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ACL degeneratio mucosa decided to undergo a surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Range of motion | At the 12 month of the follow-up
  Range of motion assessed by the means of goniometer
Range of motion | At the 24 month of the follow-up
  Range of motion assessed by the means of goniometer
Knee anterior translatory stability | At the 12 month of the follow-up
  Knee stability assessed by the means of Rollimeter-aided Lachman test - results will be presented in milimeters.
Knee anterior translatory stability | At the 24 month of the follow-up
  Knee stability assessed by the means of Rollimeter-aided Lachman test - results will be presented in milimeters.
Knee anterolateral rotational stability | At the 24 month of the follow-up
  Knee stability assessed by the means of pivot-shift test - results will be presented in grades

SECONDARY OUTCOMES:
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 12 month of the follow-up
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 24 month of the follow-up
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score (KOOS) | At the 12 month of the follow-up
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score (KOOS) | At the 24 month of the follow-up
  Min of 0 max of 100 points, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Malinowski, MD PhD, Principal Investigator — Artromedical Orthopaedic Clinic, Bełchatów, Poland
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gersing AS, Schwaiger BJ, Nevitt MC, Joseph GB, Feuerriegel G, Jungmann PM, Guimaraes JB, Facchetti L, McCulloch CE, Makowski MR, Link TM. Anterior cruciate ligament abnormalities are associated with accelerated progression of knee joint degeneration in knees with and without structural knee joint abnormalities: 96-month data from the Osteoarthritis Initiative. Osteoarthritis Cartilage. 2021 Jul;29(7):995-1005. doi: 10.1016/j.joca.2021.03.011. Epub 2021 Mar 26. PMID 33775919
- [Background] Lintz F, Pujol N, Boisrenoult P, Bargoin K, Beaufils P, Dejour D. Anterior cruciate ligament mucoid degeneration: a review of the literature and management guidelines. Knee Surg Sports Traumatol Arthrosc. 2011 Aug;19(8):1326-33. doi: 10.1007/s00167-011-1433-0. Epub 2011 Feb 18. PMID 21331652
- [Background] Sweed T, Mussa M, El-Bakoury A, Geutjens G, Metcalfe A. Management of mucoid degeneration of the anterior cruciate ligament: a systematic review. Knee Surg Relat Res. 2021 Aug 21;33(1):26. doi: 10.1186/s43019-021-00110-6. PMID 34419162
- [Background] Lee JW, Ahn JT, Gwak HG, Lee SH. Clinical Outcomes of Arthroscopic Notchplasty and Partial Resection for Mucoid Degeneration of the Anterior Cruciate Ligament. J Clin Med. 2021 Jan 16;10(2):315. doi: 10.3390/jcm10020315. PMID 33467062